CLINICAL TRIAL: NCT04279535
Title: Topical Ascorbic Acid for Treatment of Basal Cell Carcinoma
Brief Title: Topical Vitamin C for Treatment of Basal Cell Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Center for Biomedical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCC-001
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ascorbic acid (Experimental): Participants applied topical solution of ascorbic acid twice daily for 8 weeks
  Interventions: Drug: Topical Ascorbic Acid
- Imiquimod (Active Comparator): Participants applied 5% imiquimod cream topically 5x/week
  Interventions: Drug: Topical Ascorbic Acid

INTERVENTIONS:
Drug: Topical Ascorbic Acid — Twice daily application of 300 microliters of 30% ascorbic acid solution with a small cuticle brush.

SUMMARY:
Randomized coomparative trial of a 30% solution of ascorbic acid in 95% dimethylsulfoxide applied topically twice a day for 8 weeks vs 5% imiquimod cream in the treatment biopsy proven basal cell carcinomas inotherwise healthy adult patients. Outcome measure was biopsy proven resolution of the carcinoma.

DETAILED DESCRIPTION:
Importance

Skin cancer is the most common cancer in the United States, with more people diagnosed each year than all other cancers combined (1). Basal cell cancer is the most common form with an estimated 4.3 million cases diagnosed annually (2,3). Costs of treating this cancer in the U.S. are estimated at $4.8 billion annually (4). Task force consensus guidelines suggest Mohs surgery as the treatment of choice, and as the single most precise and effective treatment method (5). However, cost and issues of cosmesis are principal disadvantages.

Objective

To evaluate efficacy of a therapeutic regimen in treating basal cell cancer, consisting of 30% ascorbic acid in 95% dimethylsulfoxide topically applied at home by patients twice a day for 8 weeks, vs 5% imiquimod cream which is an FDA approved treatment for BCC.

Design, Setting, and Participants This study was carried out in accordance with principles of the Declaration of Helsinki. Detailed informed consent was obtained from each patient.

Eligible participants of any age had histologically confirmed primary, previously untreated, nodular or superficial BCC not arising at sites of high risk for sub clinical tumor spread (the nose, ear, eyelid, eyebrow, or temple ( )). Patients with infiltrative, recurrent, or morphoeic BCC were excluded from the study. Imiquimod was applied once daily for 5 days per week as per manufacturer instructions for treatment of BCC. Patients were randomly assigned to treatment group. Participants and outcome assessors were blinded to treatment protocol. Patients were seen at initial visit, 4 weeks, 8 weeks, and six weeks after treatment conclusion for final biopsy. Those participants in the IMQ group who continued through 12 weeks of treatment were seen for an additional visit. The AA treatment was a solution while the IMQ a cream, however participants were simply told they would be receiving a topical treatment with instructions on how to apply, thus the blinding remained intact.

Histopathology showed 21 nodular and 8 superficial BCC subtypes upon enrollment. Thirteen patients (8 female 5 male) with a total of 15 lesions were randomized to the ascorbic acid (AA) treatment group, and 12 patients (6 female 6 male) with 14 lesions were randomized to the imiquimod group (IMQ). There was no difference in mean size of BCC in each group ( 11.4 +/-2.1 mm vs. 13.1 +/- 1.9mm). The AA group had 11 nodular and 4 superficial BCC and the IMQ group 10 nodular and 4 superficial.

Histopathology was confirmed by 2mm partial punch biopsy leaving

the bulk of the BCC intact prior to treatment. Patients in the AA group were treated

twice daily 7 days per week with a topical solution of 30% (w/v) ascorbic acid solution in 95% (v/v) dimethylsulfoxide (DMSO) and

5% (v/v) distilled water, while the IMQ patients received twice daily application of a commercial 5% cream 5 days per week according to manufacturer recommendations for treatment of BCC. Application was made with a small cuticle brush in the AA group. Patient compliance was high and no

patient had difficulty with the application. Volume of the ascorbic acid solution applied was 0.2-0.3ml per application. Treatment was

continued for 8 wks or until the lesion cleared. Subjects in the IMQ group whose lesions had failed to resolve at 8 weeks were treated for an additional 4 weeks in conformity with reports showing better outcomes with 12 weeks of treatment with IMQ ( ).

All patients had an appointment set for Mohs surgery

after study enrollment, so in the event of treatment failure no further delay in definitive treatment would occur.

Repeat 2mm punch biopsy of each site was taken at the conclusion of the study. Patients were seen in follow up after

12, 24, and 30 months

Interventions

An 8 wk therapeutic regimen of topical 30% (w/v) ascorbic acid, 95% (v/v) dimethylsulfoxide, and 5% (v/v) distilled water applied twice daily at home, or 5% imiquimod cream applied 5/wk according to manufacturer recommendations for treating BCC.

Main Outcomes and Measures

Number of lesions out that were cancer free after 8 wks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of biopsy proven basal cell carcinoma

Exclusion Criteria:

* Absence of basal cell carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Lesion Resolution | 8 weeks
  Number of lesions resolved out of total of 6 treated.

CONTACTS AND LOCATIONS:
Overall Officials: Briant Burke, MD, Principal Investigator — CBR,Inc.
Locations (1):
- Center for Biomedical Research,Inc., Boise, Idaho, United States